CLINICAL TRIAL: NCT05378048
Title: Patient-derived-organoid (PDO) Guided Versus Conventional Therapy for Advanced Inoperable Abdominal Tumors: a Multicenter Open-label, Proof of Concept, Phase 2 Randomised Controlled Trial
Brief Title: Patient-derived-organoid (PDO) Guided Versus Conventional Therapy for Advanced Inoperable Abdominal Tumors
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: no funding support
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, James Yun-wong Lau, professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PDO
Record Dates: First submitted 2022-05-12; First posted 2022-05-17 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Organoids
Keywords: Organoids
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: patients are randomized to PDO-guided treatment or standard of care.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PDO-guided treatment (Experimental): A biopsy of the tumour will be performed for PDO culture and Genome-guided drug screening.
  An Multidisciplanary Tumour Board will review the drug screen results and recommend the use of a drug with a response in a PDO.
  Interventions: Drug: PDO-guided treatment
- standard of care (Experimental): the standard of care will include all treatments that have been reported to improve survival or quality of life in randomized trials.
  Interventions: Drug: standard of care

INTERVENTIONS:
Drug: PDO-guided treatment — A biopsy of the tumour will be performed for PDO culture and Genome-guided drug screening.
  An Multidisciplanary Tumour Board will review the drug screen results and recommend the use of a drug with a response in a PDO.
  Arms: PDO-guided treatment
Drug: standard of care — the standard of care will include all treatments that have been reported to improve survival or quality of life in randomized trials.
  Arms: standard of care

SUMMARY:
Recent studies that ex vivo drug responses on PDO models across different solid tumours can predict treatment responses to chemotherapeutic agents. In patients with metastatic or inoperable solid abdominal tumours, we perform a PDO based drug screen and to identify drugs that will confer clinical response and compared to conventional treatments

DETAILED DESCRIPTION:
Precision oncology aims to improve the clinical outcomes of patients by offering personalized treatment through identifying druggable genomic aberrations within their tumours. However, current challenges in cancer treatment have hampered the broad clinical utility of the gene-drug associations in the clinic. This is particularly valid when it comes to offering alternative treatment options for advanced inoperable patients with chemo-refractory diseases. There is currently no reliable biomarker to predict treatment response. Patient-derived organoids (PDOs) closely resemble both pheno- and genotypically to patients' tumours. In observational studies, anticancer drug screening ex vivo on PDOs has been shown to predict clinical response with high sensitivity and specificity. PDO-based drug screen represents a truly personalised platform by predicting patient-specific drug response with high accuracy. Recent technical advancements in growing these PDO 'avatars' from biopsies have made it possible to find anticancer drug options in tumours from advanced inoperable patients, and explore new possibilities for treatment options that otherwise would be missed by standard conventional therapies. PDO-based drug assays permit examination of combinatorial drug testing ex vivo and potentially offer patients treatment options. The clinical utility of treatment based on PDO informed drug options however has not been established. We hypothesize that treatment guided by PDO-based drug screens, when compared to conventional treatment, can lead to better treatment response and clinical outcomes. We propose a phase 2 proof-of-concept randomized controlled trial in patients with inoperable or metastatic abdominal tumours refractory to at least one chemotherapeutic agent. Our primary endpoint to this randomised trial is progression-free survival (PFS) at 12 months. In this trial, we in addition expand our current bio-resource of PDOs, and further valid PDO guided treatment model by comparing ex vivo PDO drug response to patients' clinical response.

ELIGIBILITY:
Inclusion Criteria:

* patients should be older than 18 years, able to provide written consents to trial participation, with Eastern cooperative oncology group performance status of 0 or 1, With measurable disease in accordance with response evaluation criteria in solid tumours (RECIST) version 11. [ 10 ] With a neutrophil count, hemoglobin > 9g/dl, serum creatinine <1.5 x upper limit of normal, serum bilirubin < 1.5 x normal, and aspartate and alanine aminotransferases (<3 x ULN or <5x in those with liver metastasis) Ejection Fraction >50% of normal. The disease is accessible for a biopsy (radiologic or endoscopic) or resection of a metastatic site.

Exclusion Criteria:

* unable to give consent, could not obtain a biopsy

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-07-04 (Estimated); Primary Completion 2025-07-03 (Estimated); Study Completion 2025-07-03 (Estimated)

PRIMARY OUTCOMES:
Tumor progression-free survival | 12 months after randomization
  The length of time after patients have received treatment and have no detectable disease and have no detectable disease

SECONDARY OUTCOMES:
the rate of overall survival | 12 months after randomization
  the percentage of people who are alive
tumour response rates | 12 months after randomization
  the assessment of the tumor burden (TB) after the treatment
rate of successful organoid culture and drug screen organoid culture | 4-6 weeks after culture
  the percentage of survival organoid and the availability of at least one drug to which PDO responds
rate of serious adverse events | 12 months after randomization
  the rate of side effects of drug, prolonging the hospitalization

CONTACTS AND LOCATIONS:
Locations (1):
- Department of surgery , Prince of Wales Hospital, Hong Kong, N.T., Hong Kong

IPD SHARING:
Plan to Share IPD: No